CLINICAL TRIAL: NCT01579357
Title: Pharmacokinetics and Metabolic Activation of Capecitabine When Given Concomitantly With Oxaliplatin and the Monoclonal Antibody Cetuximab
Brief Title: Pharmacokinetics and Metabolic Activation of Capecitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AGMT-Capecet_PK
Record Dates: First submitted 2012-03-29; First posted 2012-04-18 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal carcinoma; K-ras wild type; Capecitabine; Cetuximab; Oxaliplatin; Pharmacokinetics; exclude a possible influence of CETUX; plasma disposition; metabolic activation; CCB; OxPt
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Capecitabine in week 1,2,4,5,7 and 8 Cetuximab in week 3 to 9 Oxaliplatin in week 7
  Interventions: Other: blood samples
- B (Other): Capecitabine in weeks 1,2,4,5,7, and 8 Cetuximab in weeks 1,8 and 9 Oxaliplatin in week 7
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — Draw blood samples in week 1 (day 1 and day 5), in week 4 (day 1 and day 5) and in week 7 (day 1 and day 5).
  day 1: pre dose, 30,60,90,120,150,180,240,300 and 360min day 5: pre dose, 30,60,90,120min

SUMMARY:
The objective of this pharmacokinetic study is to exclude a possible influence of CETUX on the plasma disposition and metabolic activation of Capecitabine (CCB) and when this regimen is given combined with Oxaliplatin (OxPt).

ELIGIBILITY:
Inclusion Criteria selected:

* signed written informed consent
* male or female > 18 years
* K-ras wild type adenocarcinoma of the colon or rectum
* metastatic colorectal carcinoma
* ECOG <= 2

Exclusion Criteria selected:

* brain metastasis
* previous chemotherapy
* stage 3 or 4 heart failure
* uncontrolled angina
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Influence of Cetuximab on metabolic activation of Capecitabine | 9 weeks
  Curve fitting of drug and metabolite concentrations will be performed. For pharmacokinetic modelling of CCB and metabolites, a non-compartment model for extravascular input will be used. For calculation of AUC and AUMC the linear trapezoid rule will be applied for the ascending part of the concentraion-time curve and the log-linear trapezoidal rule for the descending part of the concentration-time curve.

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - PMU Salzburg, Salzburg, Salzburg
  - AKH Wien, Vienna, Vienna
  - Kaiser Franz Josef Spital, Vienna, Vienna

REFERENCES:
- See also: Sponsor — http://www.agmt.at